CLINICAL TRIAL: NCT05066958
Title: Safety and Efficacy Study of an Ex-vivo Antigen-primed Donor Memory Lymphocyte Infusion for the Enhancement of Immunity to Viral Infections Among Recipients of Allogeneic Hematopoietic Stem Cell Transplantation on the Platform of Selective Immunomagnetic Depletion of T-lymphocytes
Brief Title: Ex-vivo Primed Memory Donor Lymphocyte Infusion to Boost Anti-viral Immunity After T-cell Depleted HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCPHOI-2020-06
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia; High Risk Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia, in Relapse; High Risk Acute Lymphoblastic Leukemia; Acute Biphenotypic Leukemia in Relapse; Non-hodgkin Lymphoma; Myelodysplastic Syndromes
Keywords: Hematopoietic stem cell transplantation; alpha/beta T cell depletion; CD45RA depletion; immune reconstitution; viral infections; ELISPOT
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Virus Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- boost anti-viral immunity after T-cell depleted HSCT (Experimental)
  Interventions: Biological: boost anti-viral immunity after T-cell depleted HSCT

INTERVENTIONS:
Biological: boost anti-viral immunity after T-cell depleted HSCT — * Registration and informed consent sign
  * Screening clinical and laboratory examination, assessment of compliance with inclusion criteria
  * Survey of the recipient and potential donors
  * Donor selection
  * The study of the immune response to relevant antigens in the donor and recipient
  * Pre-transplant conditioning
  * Stimulation of the donor and apheresis of peripheral blood mononuclear cells
  * Graft processing
  * The manufacturing of cell product
  * Transplant Infusion
  * Antigen-primed memory DLI infusion
  * Inpatient care until day +30
  * Outpatient monitoring and screening

SUMMARY:
HSCT from an allogeneic donor is the standard therapy for high-risk hematopoietic malignancies and a wide range of severe non-malignant diseases of the blood and immune system. The possibility of performing HSCT was significantly limited by the availability of donors compatible with the MHC system. However, modern ex-vivo and in vivo technologies for depletion of T lymphocytes have made it possible to improve the outcomes of HSCT from partially compatible related (haploidentical) donors. In representative groups, it was shown that the success of HSCT from haploidentical donors is not inferior to standard procedures of HSCT from HLA-compatible unrelated donors. HSCT from haploidentical donors in children associated with the deficit of the adaptive immune response, which persists up to 6 months after HSCT and can be an increased risk of death of the patient from opportunistic infections. To solve this problem, the method of infusion of low doses of donor memory T lymphocytes was introduced. This technology is based on the possibility of adoptive transfer of memory immune response to key viral pathogens from donor to recipient. Such infusions have been shown to be safe and to accelerate the recovery of the pathogen-specific immune response. The expansion of virus-specific T lymphocytes in the recipient's body depends on exposure to the relevant antigen in vivo. Thus, in the absence of contact with the viral antigen, the adoptive transfer of memory T lymphocytes is not accompanied in vivo by the expansion of virus-specific lymphocytes and does not form a circulating pool of memory T lymphocytes, that can protect the patient from infections. Therefore the investigators assume that ex-vivo priming of donor memory lymphocytes with relevant antigens can provide optimal antigenic stimulation and may solve the problem of restoring immunological reactivity in the early stages after HSCT. Technically ex-vivo primed memory T lymphocytes will be generated by short incubation of CD45RA-depleted fraction of the graft (a product of T lymphocyte depletion) with a pool of GMP-quality peptides representing a number of key proteins of the viral pathogens. The following are proposed as targeted antigens: CMV pp65, EBV EBNA-1, EBV LMP12A, Adeno AdV5 Hexon, BKV LT, BKV VP1. An infusion of donor memory lymphocytes will be performed on the day +1 after transplantation. Parameters of the assessment will be safety and efficacy (immune response by day 60 and stability (responses by day 180).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the patient (ages 14 to 18) and / or his legal representative (ages 0 to 18).
2. The patient has an indication for allogeneic transplantation of hematopoietic stem cells established in accordance with the current regulatory framework
3. Planned HSCT selective immunomagnetic depletion of alpha/betta T lymphocytes
4. Karnovsky or Lansky index more than 50%
5. Life expectancy at least 4 weeks
6. Heart function: ejection fraction of at least 40%
7. Consent to continue follow-up for 5 years

Exclusion Criteria:

1. Acute viral hepatitis or acute HIV infection
2. Hypoxemia with SaO2 <90%
3. Bilirubin> 3 norms
4. Creatinine> 3 norms
5. Pregnancy and lactation
6. Severe uncontrolled infection
7. Severe (>?) pathology of the central nervous system (epilepsy, dementia, organic damage to the central nervous system, psychosis)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
acute Graft Versus Host Disease | 100 days after HSCT
  Cumulative risk of developing of acute Graft Versus Host Disease (aGVHD) (evaluation period is 100 days) stage II-IV
The proportion of patients with detectable T-cell response (IFNgamma ELISPOT) to CMV | after HSCT by day + 30 and by day + 180
  The proportion of patients with detectable peripheral blood T-lymphocytes specific for CMV antigens
The proportion of patients with detectable T-cell response (IFNgamma ELISPOT) to ADV | after HSCT by day + 30 and by day + 180
  The proportion of patients with detectable peripheral blood T-lymphocytes specific for ADV antigens
The proportion of patients with detectable T-cell response (IFNgamma ELISPOT) to EBV | after HSCT by day + 30 and by day + 180
  The proportion of patients with detectable peripheral blood T-lymphocytes specific for EBV antigens

SECONDARY OUTCOMES:
Cumulative Incidence of developing chronic GVHD | after HSCT up to 2 years
  Cumulative Incidence of developing chronic GVHD
Cumulative Incidence of recurrence of leukemia CI of relapse | after HSCT up to 2 years
  Cumulative Incidence of recurrence of leukemia
TRM | after HSCT up to 2 years
  Cumulative Incidence of transplant-related mortality
OS | after HSCT up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mikchail m Maschan, Study Director — Chief HSCT department at Federal Research Center for pediatric hematology, oncology and immunology
Locations (1):
- Federal Research Center for pediatric hematology, oncology and immunology, Moscow, Russia